CLINICAL TRIAL: NCT02673528
Title: Laparoscopic Assisted or Total Laparoscopic Appendectomy in Patients With Uncomplicated Acute Appendicitis: a Matched Case-control, Cost-utility Study
Brief Title: Laparoscopic Assisted or Total Laparoscopic Appendectomy
Status: Completed | Type: Observational
Sponsor: Medical Park Gaziantep Hospital (Other)
Collaborators: Bahçeşehir University (Other); Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Mehmet Kaplan, Head of General Surgery, Medical Park Gaziantep Hospital
Other Study IDs: MK-007-LAA
Record Dates: First submitted 2016-01-21; First posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Acute Appendicitis
Keywords: appendectomy; laparoscopy; laparoscopic assisted appendectomy; cost utility
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — appendectomy material
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Directly underwent TLA: Patients with the diagnosis who underwent directly total laparoscopic appendectomy
  Interventions: Procedure: Laparoscopic appendectomy
- Lap Assisted App: Patients with the diagnosis of acute appendicitis who underwent a successful laparoscopic assisted appendectomy
  Interventions: Procedure: Laparoscopic appendectomy
- Advanced to TLA: Patients with the diagnosis of acute appendicitis in whom laparoscopic assisted appendectomy attempted; however, because it fail advanced to total laparoscopic appendectomy.
  Interventions: Procedure: Laparoscopic appendectomy

INTERVENTIONS:
Procedure: Laparoscopic appendectomy — Two types of laparoscopic surgery were performed. Total laparoscopic appendectomy or laparoscopic assisted appendectomy
  Other Names: laparoscopic assisted appendectomy

SUMMARY:
Acute appendicitis (AA), is a common intra-abdominal surgical pathology with the overall incidence of approximately 7% and mortality of 0.2-0.8%. Treatment of choice is the surgical removal of the inflamed appendix by using open or laparoscopic appendectomy.

Following laparoscopic appendectomy (LA) proved to be a feasible and at least as safe as the corresponding open procedure, it has rapidly gained worldwide acceptance. The traditional approach to LA uses three ports. Over the past decade, successful attempts to perform the procedure with fewer ports have been reported.

The authors' primary objectives were to 1) identify a simple, safe and feasible way to perform laparoscopic appendectomy in patients with uncomplicated acute appendicitis. 2) determine the health related quality of life of the patients and calculate the cost per quality adjusted life years (QALYs) gained after the procedures (LAA and TLA). 3) Purpose a surgical algorithm when approaching to acute appendicitis with the consideration of quality of health and cost.

DETAILED DESCRIPTION:
Acute appendicitis (AA), is a common intra-abdominal surgical pathology with the overall incidence of approximately 7% and mortality of 0.2-0.8%. Treatment of choice is the surgical removal of the inflamed appendix by using open or laparoscopic appendectomy. Until the first laparoscopic removal of an inflamed appendix by Kurt Semm in 1980, the gold standard for surgical treatment of acute appendicitis remained open appendectomy as first described by McBurney in 1891.

At the beginning, LA remained questionable whether the benefits of the procedure outweigh over its disadvantages. However, since laparoscopic technology advances and surgeons' expertise increases, many surgeons have successfully performed a multitude of laparoscopic procedures for AA, with a continued increasing trend in its use. Eventually, after LA proved to be a feasible and at least as safe as the corresponding open procedure, it has rapidly gained worldwide acceptance.

There are more techniques for LA in the literature but only a few of them have gained to access and described in modern textbooks. The traditional approach to LA uses three ports. Over the past decade, successful attempts to perform the procedure with fewer ports have been reported which include two-port techniques, single-port techniques, and hybrid approaches. The two-port appendectomy technique consist of one port providing access for a rigid telescope with a working channel, and second port for a grasping forceps that is used to retract the appendix. In the single-port assisted technique, after a stitch is placed between the appendix and the anterior abdominal wall to pull the appendix and create a tension to facilitate dissection, and then appendectomy is performed intracorporeally. The hybrid technique formed from the combination of both open and laparoscopic approaches. Namely the appendix is pulled out through the only or one of the port, and a traditional open appendectomy is then performed extracorporeally.

The authors' primary objectives were to 1) identify a simple, safe and feasible way to perform laparoscopic appendectomy in patients with uncomplicated acute appendicitis. 2) determine the health related quality of life of the patients using Euro Qol (EQ) - 5 Dimensions (5D) - 3 Levels (3L) (EQ-5D-3L) and Visual Analogue Scale (VAS) and calculate the cost per quality adjusted life years (QALYs) gained after the procedures (LAA and TLA). 3) Purpose a surgical algorithm when approaching to acute appendicitis with the consideration of quality of health and cost. For these purposes, a case-control study was designed in January 2015 to investigate these issues.

ELIGIBILITY:
Inclusion Criteria:

* all acute appendicitis patients underwent total laparoscopic appendectomy or laparoscopic assisted appendectomy

Exclusion Criteria:

* no written informed consent

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The control group (Group 1) comprised 108 matched-cases of uncomplicated appendicitis operated with total laparoscopic appendectomy within the period January 2008 through July 2011.
  The study group (Group 2) is represented by 108 consecutive patients diagnosed with uncomplicated acute appendicitis, operated with lap assisted appendectomy.
  Group 3 consisted of 211 patients with uncomplicated appendicitis, in whom Lap assisted ap were unsuccessful because of several reasons, were underwent to Total Lap App within the same period
Sampling Method: Probability Sample
Enrollment: 451 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
A weekly change in EQ-5D-3L scores (Euro Qol 5 dimensions 3 levels) | two times: 7th and 14th day after the surgery
  health related evaluation
A weekly change in EQ-VAS scores (Euro Qol Visual Analogue Scale) | two times: 7th and 14th day after the surgery
  visual analogue scale of health related evaluation
Calculation of Cost utility | within 1 month after surgery
  depends on the calculation of hospital based costs and QALY

SECONDARY OUTCOMES:
Ratio of conversion to TLA | within the first month after completion of the patient recruitment
  Ratio of conversion of laparoscopic assisted to total laparoscopic appendectomy
Mean BMI of patients in the groups | within 1 month after completion of the patient recruitment
  to asses the effect of higher body mass index on the success of procedures the authors will calculate BMI in each group
The rate of the location of appendix | within 1 month after completion of the patient recruitment
  To asses the the effect of the location of the appendix on the preference of surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Kaplan, M.D., Study Director — Bahçeşehir Üniversitesi Tıp Fakültesi

IPD SHARING:
Plan to Share IPD: No